CLINICAL TRIAL: NCT04337177
Title: Pilot Pharmacokinetic Study of VAL-413 (Orotecan®) in Patients With Recurrent Pediatric Solid Tumors
Brief Title: Flavored, Oral Irinotecan VAL-413 (Orotecan®) Given With Temozolomide for Treatment of Recurrent Pediatric Solid Tumors
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Valent Technologies, LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: VAL-10-001
Record Dates: First submitted 2020-03-30; First posted 2020-04-07 (Actual); Last update posted 2025-09-23 (Actual); Status verified 2025-09

CONDITIONS: Solid Tumors; Neuroblastoma; Rhabdomyosarcoma; Ewing Sarcoma; Hepatoblastoma; Medulloblastoma
Keywords: irinotecan; pediatric; solid tumor; neuroblastoma; rhabdomyosarcoma; Ewing sarcoma; hepatoblastoma; medulloblastoma; recurrent
MeSH Terms: conditions — Neuroblastoma; Rhabdomyosarcoma; Sarcoma, Ewing; Hepatoblastoma; Medulloblastoma; Recurrence | interventions — Temozolomide

STUDY DESIGN:
Intervention Model Description: Two different dose levels of VAL-413 (Orotecan®) will be studied in combination with fixed-dose temozolomide using a standard 3 + 3 phase I design. The first three patients will receive temozolomide in combination with Orotecan® at 90 mg/m2/day, which is the standard dose of irinotecan. If no dose-limiting toxicity (DLT) occurs during Cycle 1 in these patients, then subsequent patients will start Cycle 1 using a Orotecan® dose of 110 mg/m2/day. In the event the starting dose of 90 mg/m2/day is not tolerable due to toxicity, a lower starting dose of 75 mg/m2/day may be implemented.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- 90 mg/m2/day VAL-413 (Orotecan®) (Experimental): Orotecan® at 90 mg/m2/day administered with Temozolomide at 100 mg/m2/day orally for 5 consecutive days at the beginning of every 21-day cycle. A single dose of the intravenous preparation of irinotecan taken orally (IRN-IVPO) will be substituted at the same dosage as Orotecan® for during Cycle 1.
  Interventions: Drug: VAL-413; Drug: Temozolomide
- 110 mg/m2/day VAL-413 (Orotecan®) (Experimental): Orotecan® at 110 mg/m2/day administered with Temozolomide at 100 mg/m2/day orally for 5 consecutive days at the beginning of every 21-day cycle. A single dose of the intravenous preparation of irinotecan taken orally (IRN-IVPO) will be substituted at the same dosage as Orotecan® for during Cycle 1.
  Interventions: Drug: VAL-413; Drug: Temozolomide
- 75 mg/m2/day VAL-413 (Orotecan®) (Experimental): In the event the 90 mg/m2/day starting dose is not tolerable due to toxicity, a lower starting dose of 75 mg/m2/day may be implemented. Orotecan® at 75 mg/m2/day administered with Temozolomide at 100 mg/m2/day orally for 5 consecutive days at the beginning of every 21-day cycle. A single dose of the intravenous preparation of irinotecan taken orally (IRN-IVPO) will be substituted at the same dosage as Orotecan® for during Cycle 1.
  Interventions: Drug: VAL-413; Drug: Temozolomide

INTERVENTIONS:
Drug: VAL-413 — a flavored preparation of orally administered irinotecan
  Other Names: Orotecan®
Drug: Temozolomide — alkylating oral chemotherapy agent used to treatment brain cancers
  Other Names: Temodar; Temodal; Temcad; TMZ

SUMMARY:
A pilot pharmacokinetic trial to determine the safety and efficacy of a flavored, orally administered irinotecan VAL-413 (Orotecan®) given with temozolomide for treatment of recurrent pediatric solid tumors including but not limited to neuroblastoma, rhabdomyosarcoma, Ewing sarcoma, hepatoblastoma and medulloblastoma

DETAILED DESCRIPTION:
Up to 20 patients ≥ 1 year of age or ≤ 30 years of age with recurrent pediatric solid tumors will be enrolled. During the first cycle of treatment, each patient will receive 4 daily doses of VAL-413 (Orotecan®) and one daily dose of the intravenous preparation of irinotecan taken orally (IRN-IVPO), together with 5 days of concurrent temozolomide. During all subsequent cycles, only Orotecan® will be given with temozolomide in 5 day courses administered every 21 days as tolerated.

The dosing regimen in this study will be Temozolomide at 100 mg/m2/day with Orotecan® at either 90 or 110mg/m2/day, administered orally for 5 consecutive days at the beginning of every 21-day cycle. A single dose of IRN-IVPO will be substituted at the same dosage as Orotecan® during Cycle 1. Up to 17 cycles of treatment may be administered on this study.

Data collected from this study will allow for an assessment of Orotecan® safety and efficacy. Interval medical histories, targeted physical exams, complete blood counts, and other laboratory and safety assessments will be performed at Day 1 of each treatment cycle for all study subjects. At baseline and during study, disease status will be assessed by appropriate clinical and imaging evaluation (CT, MRI, or PET) and using Response Evaluation Criteria in Solid Tumors (RECIST), International Neuroblastoma Response Criteria (INRC) for patients with neuroblastoma, or the Children's Oncology Group Response Criteria for CNS tumors. In addition, a single-response taste survey will be conducted on Day 1 and Day 4 of the first cycle, which will allow patients to evaluate the taste of Orotecan®. Serum samples will be collected at various time points on Days 1 and 4 during Cycle 1 to characterize and compare the pharmacokinetic profiles of Orotecan® and conventional irinotecan given orally.

Assessment of first-cycle toxicity will be used to identify the recommended phase II dose for Orotecan®. Toxicity will be evaluated and documented using NCI CTCAE guidelines. The recommended Phase II dose will be identified as the highest dose at which no more than 1 of 6 patients experiences a first cycle dose limiting toxicity (DLT). Additional study subjects may be enrolled at the recommended Phase II dose to ensure balanced safety and pharmacokinetic data is obtained for at least 3 patients < 12 years old and at least 3 patients > 12 years old.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must be 1 year of age to ≤ 30 years of age at the time of study entry.
2. Patients must have had histologic verification of a solid tumor or CNS tumor at either original diagnosis or relapse.
3. Measurable or evaluable disease is not required for enrollment on this safety/feasibility study.
4. Patient's current disease state must be one for which there is no known curative therapy or therapy proven to prolong survival with an acceptable quality of life or for which irinotecan and/or temozolomide are acceptable therapeutic options based on existing standard of care available.
5. Karnofsky Performance Status ≥ 50% for patients > 16 years of age and Lansky Performance Status ≥ 50 for patients ≤ 16 years of age. Patients who are unable to walk because of paralysis, but who are up in a wheelchair, will be considered ambulatory for the purpose of assessing the performance score.
6. Males or females of reproductive potential may not participate unless they have agreed to use an effective contraception method during and for 30 days after study treatment. (Abstinence is considered an acceptable method of effective contraception.)
7. Prior treatment with temozolomide, vincristine or irinotecan is allowed, although patients must not have had disease progression while receiving either irinotecan, vincristine or temozolomide.
8. Patients must have recovered from the acute toxic effects of all prior chemotherapy, immunotherapy, or radiotherapy prior to entering this study, as described below:

   1. Myelosuppressive chemotherapy: patients must not have received myelosuppressive chemotherapy within 21 days of first study treatment, but nitrosourea within 8 weeks (42 days) of first study treatment
   2. Anti-cancer agents not known to be myelosuppressive (e.g., not associated with drops in platelet or neutrophil count): must not have received these therapies within 7 days of first study treatment, or at least 5 half-lives of the agent (whichever is longer)
   3. Antibody therapy: At least 4 weeks must have elapsed since last antibody dose prior to first study treatment
   4. Radiation therapy: At least two weeks must have elapsed since last local palliative radiation (small port) prior to first study treatment. At least 6 weeks must have elapsed if more substantial radiation was administered (e.g., >50% pelvis, craniospinal, whole body), or therapeutic radiolabeled 131I MIBG or other radiopharmaceutical therapy.
   5. High-Dose Chemotherapy with Autologous Stem Cell Transplant/Rescue: At least two months must have elapsed since receiving autologous hematopoietic stem cells prior to first study treatment. Patients who have had allogeneic transplants are ineligible.
   6. Hematopoietic growth factors: must not have been received in the 14 days prior to first study treatment for a long-acting growth factor (e.g., pegfilgrastim), or 7 days prior to first study treatment for short-acting growth factor.
9. Peripheral absolute neutrophil count (ANC) ≥ 1,000/µL
10. Platelet count ≥100,000/µL (transfusion independent, defined as not receiving platelet transfusions within a 7-day period prior to first study treatment)
11. Hemoglobin ≥ 8.0 gm/dL (may receive RBC transfusions) NOTE: Patients with metastatic tumor in the bone marrow ARE eligible provided the above hematologic criteria are met.
12. Creatinine clearance or radioisotope GFR ≥ 70mL/min/1.73 m2 or Serum creatinine based on age/gender as follows:

    Age Maximum Serum Creatinine (mg/dL) Male Female 1 to < 2 years 0.6 0.6 2 to < 6 years 0.8 0.8 6 to < 10 years 1 1 10 to < 13 years 1.2 1.2 13 to < 16 years 1.5 1.4

    ≥ 16 years 1.7 1.4

    The threshold creatinine values in this Table were derived from the Schwartz formula for estimating GFR (Schwartz et al. J. Peds, 106:522, 1985) utilizing child length and stature data published by the CDC.
13. Bilirubin (sum of conjugated + unconjugated) ≤ 1.5 x upper limit of normal (ULN) for age
14. SGPT (ALT) ≤ 5 x upper limit of normal (ULN) for age
15. Serum albumin ≥ 2 g/dL

Exclusion Criteria:

1. Patients with a history of severe allergic reaction (e.g., more than simple rash) to dacarbazine or third-generation cephalosporins are ineligible.
2. Pregnant or breast-feeding women will not be entered on this study due to potential risks of fetal and teratogenic adverse events. A pregnancy test must be obtained prior to starting chemotherapy in post-menarchal female patients.
3. Patients who are currently receiving investigational drugs, or who have received an investigational drug within the last 7 days prior to first study treatment, are ineligible.
4. Patients who are currently receiving other anti-cancer agents are ineligible.
5. Patients taking strong inducers of CYP3A4, including but not limited to phenobarbital, phenytoin, carbamazepine, oxcarbazepine (Trileptal), rifampin, voriconazole, itraconazole, ketoconazole or other systemically-administered azole antifungal drugs, aprepitant (Emend) or St. John's Wort, in the 2 weeks prior to first study treatment are ineligible.
6. Patients taking strong inhibitors of CYP3A4 or UGT1A1 in the 1 week prior to first study treatment are ineligible.
7. Patients must not be receiving medications known to inhibit platelet function or known to selectively inhibit cyclooxygenase activity. Medicines in this class are excluded, with the exception of acetaminophen.
8. Patients who have uncontrolled infections, require IV antibiotics at time of enrollment, or who are currently receiving treatment for Clostridium difficile infection are excluded.
9. Patients who in the opinion of the investigator may not be able to comply with the safety monitoring requirements of the study are not eligible.

Ages: 1 Year to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 20 (Estimated)
Dates: Start 2021-10-25 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Recommended Phase II Dose (RP2D) | 17 months
  To establish the recommended Phase II dose of a flavored preparation of orally administered irinotecan VAL-413 (Orotecan®) when given in combination with temozolomide for 5 consecutive days

SECONDARY OUTCOMES:
Cmax | 1 day
  Maximum observed concentration of VAL-413 (Orotecan®) on Day 1
Tmax | 1 day
  Time of observed VAL-413 (Orotecan®) Cmax on Day 1
AUClast | 1 day
  Area under the concentration-time curve from pre-dose (time 0) to the time of the last quantifiable VAL-413 (Orotecan®) concentration on Day 1
AUCinf | 1 day
  Area under the concentration-time curve for VAL-413 (Orotecan®) extrapolated to infinity on Day 1
CL/F | 1 day
  Total oral body clearance at steady state calculated as VAL-413 (Orotecan®) dose/AUC on Day 1
MRT | 1 day
  Mean Residence Time for VAL-413 (Orotecan®) calculated as AUMC/AUC where AUMC is Area under the Moment Curve
Vz | 1 day
  The apparent volume of distribution for VAL-413 (Orotecan®) during the terminal phase
Lambda z | 1 day
  The terminal elimination rate constant determined by selection of at least three decreasing data points on the terminal phase of the concentration time curve for VAL-413 (Orotecan®) on Day 1
T1/2 | 1 day
  Terminal elimination half-life of VAL-413 (Orotecan®) on Day 1 determined from 0.693/Lambda z
Palatability | 1 month
  To evaluate the palatability of VAL-413 (Orotecan®) using a proprietary Valent Taste Survey which allows pediatric patients or their parents to rate how agreeable they find the flavor of VAL-413 (Orotecan®), on scale from 7, Like Very Much down to 1, Dislike Very Much
Adverse Events | 17 months
  To assess the toxicity profile of this combination therapy using NCI CTCAE guidelines
Treatment Response | 17 months
  To assess treatment response using the Response Evaluation Criteria in Solid Tumors (RECIST) guideline, or for patients with neuroblastoma, the International Neuroblastoma Response Criteria (INRC) guideline

CONTACTS AND LOCATIONS:
Overall Officials: Lars Wagner, M.D., Principal Investigator — Duke University Children's Hospital & Health Center; James Geller, M.D., Principal Investigator — Cincinnati Children's Hospital Medical Center (CCHMC); Meghann McManus, D.O., Principal Investigator — Sarah Cannon Research Institute, Pediatric Hematology & Oncology; Javier Oesterheld, M.D., Principal Investigator — Atrium Health Levine Children's Hospital - Carolinas Medical Center; Patrick Thompson, M.D., Principal Investigator — UNC Chapel Hill - North Carolina Cancer Hospital; Aerang Kim, M.D., Principal Investigator — Children's National Hospital - Washington, DC; Kieuhoa Vo, M.D., Principal Investigator — UCSF - Mission Bay, Benioff Children's Hospital; Kyle Jackson, M.D., Principal Investigator — Indiana University School of Medicine, Riley Hospital for Children
Locations (8):
- United States (8):
  - UCSF, Mission Bay - Benioff Children's Hospital, San Francisco, California
  - Children's National Research Institute - Children's National Hospital, Washington D.C., District of Columbia
  - Indiana University School of Medicine, Riley Hospital for Children, Indianapolis, Indiana
  - University of North Carolina at Chapel Hill - North Carolina Cancer Hospital, Chapel Hill, North Carolina
  - Atrium Health Levine Children's Hospital - Carolinas Medical Center, Charlotte, North Carolina
  - Duke University Children's Hospital and Health Center, Durham, North Carolina
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Sarah Cannon Research Institute, Pediatric Hematology & Oncology, Nashville, Tennessee

IPD SHARING:
Plan to Share IPD: No